CLINICAL TRIAL: NCT06429501
Title: The Impact of Perioperative Nerve Block on Opioid Use After Craniomaxillofacial Trauma Surgery: A Randomized Controlled Trial
Brief Title: Local Anesthesia for Facial Fractures
Acronym: LAFF
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202401085
Record Dates: First submitted 2024-04-23; First posted 2024-05-28 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Pain Management
Keywords: otolaryngology; surgery; facial plastic; trauma
MeSH Terms: conditions — Agnosia; Wounds and Injuries | interventions — Bupivacaine; Epinephrine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Double-blinded, placebo-controlled randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study team members and the participants will be blinded to the assignment of participants in the study groups. Only the pharmacist will prepare the study syringes and the unblinded statistician will have access to the study group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupivacaine injection (Experimental): The surgeon will be provided with a 10 mL syringe, and he/she will be blinded to the contents of the syringe. The appropriate landmarks will be identified, and a 21, 25, or 27- gauge needle will be used to perform the nerve block with 0.25% bupivacaine.
  Interventions: Drug: Bupivacaine/Epinephrine
- Saline injection (Placebo Comparator): The placebo sham injection will be performed in an identical fashion as the nerve block with the exception of using 10 mL of 0.9% saline injection instead of bupivacaine.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Bupivacaine/Epinephrine — injection
  Arms: Bupivacaine injection
Drug: Saline — injection
  Arms: Saline injection

SUMMARY:
The study is a double-blind randomized, placebo controlled trial examining the impact of perioperative bupivacaine nerve block on PACU recovery metrics. Patients with operative facial fractures are randomized to receive either bupivacaine or saline injections prior to the anesthesia emergence.

DETAILED DESCRIPTION:
Effective pain management is critical to successful postoperative care and is known to decrease patient morbidity, incurred patient and hospital costs, and length of hospital stay. Pain and nausea after surgery for traumatic facial fractures can limit patients' early morbidity, oral intake, and ability to communicate.

The study is a double-blind randomized, placebo controlled trial examining the impact of perioperative bupivacaine nerve block on PACU recovery metrics. Patients with operative mandibular or midface fractures are randomized to receive either bupivacaine or saline injections prior to the anesthesia emergence. The primary outcome measure is the amount of opioid that patients receive in PACU in morphine milligram equivalent (MMEs).

The purpose of the study is to define whether a perioperative bupivacaine nerve block results in a decrease in the amounts of opioids and antiemetics that patients receive in PACU after CMF trauma surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18 and over
2. Isolated facial fracture to the mandible and/or midface undergoing surgical repair
3. No allergy to local anesthetic
4. Ability to read, write, and understand English

Exclusion Criteria:

1. Patients under the age of 18
2. Isolated nasal bone fracture
3. Polytrauma (I.e. injury pattern resulting in hospital admission for multiple bony fractures outside of the face)
4. Allergy to local anesthetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Impact of a perioperative bupivacaine nerve block on PACU opioid use as assessed by the amount of opioids received in morphine milligram equivalents (MMEs). | day 1 or the day of surgery
  To evaluate the impact of a perioperative bupivacaine nerve block on PACU opioid use in patients undergoing operative fixation of facial fractures compared to placebo nerve block assessment of the amount of opioids that patients receive in PACU in morphine milligram equivalents (MMEs) will be calculated.

SECONDARY OUTCOMES:
Impact of a perioperative bupivacaine nerve block on antiemetic use as assessed by the numbers who receive opioids and antiemetics, amount of antiemetics, pain score, frequency of emesis, and time until discharge. | within 1 month post surgery
  To evaluate the impact of a perioperative bupivacaine nerve block on PACU antiemetic use in patients undergoing operative fixation of facial fractures compared to placebo nerve block. Additional variables that will be collected perioperatively include the medications used for induction/maintenance of anesthesia as well as intraoperative analgesia (I.e. fentanyl, hydromorphone, morphine, acetaminophen, ketorolac, etc.), operative time, estimated blood loss, and intraoperative complications.

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Hari_Raj, MD, Principal Investigator — Washington University School of Medicine; Jay Piccirillo, MD, Study Director — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hedegaard H, Minino AM, Spencer MR, Warner M. Drug Overdose Deaths in the United States, 1999-2020. NCHS Data Brief. 2021 Dec;(426):1-8. PMID 34978529
- [Background] Abraham AJ, Rieckmann T, Gu Y, Lind BK. Inappropriate Opioid Prescribing in Oregon's Coordinated Care Organizations. J Addict Med. 2020 Jul/Aug;14(4):293-299. doi: 10.1097/ADM.0000000000000569. PMID 31609864
- [Background] BJC Healthcare. Level I Trauma Center. Barnes-Jewish Hospital. https://www.barnesjewish.org/Medical-Services/Trauma-Acute-CareSurgery/Level-I-Trauma-Center
- [Background] Lapidus JB, Santosa KB, Skolnick GB, Som A, Cho GJ, Waljee JF, AuBuchon JD, Patel KB. Opioid Prescribing and Use Patterns in Postsurgical Facial Trauma Patients. Plast Reconstr Surg. 2020 Mar;145(3):780-789. doi: 10.1097/PRS.0000000000006588. PMID 32097326
- [Background] Perloff MD, Chung JS. Urgent care peripheral nerve blocks for refractory trigeminal neuralgia. Am J Emerg Med. 2018 Nov;36(11):2058-2060. doi: 10.1016/j.ajem.2018.08.019. Epub 2018 Aug 8. PMID 30119988
- [Background] Staity G, Saadi RA, Pool C, Lighthall JG. The Safety Profile of Liposomal Bupivacaine Use in Septorhinoplasty. Facial Plast Surg Aesthet Med. 2022 May-Jun;24(3):202-206. doi: 10.1089/fpsam.2020.0544. Epub 2021 Feb 22. PMID 33617355
- [Background] Schumacher JK, Cristel RT, Talugula S, Shah AR. The Use of Adjunctive Perioperative Nerve Blocks in Rhinoplasty in the Immediate Postoperative Period. Facial Plast Surg Aesthet Med. 2023 Jul-Aug;25(4):361-362. doi: 10.1089/fpsam.2022.0125. Epub 2022 Sep 14. No abstract available. PMID 36106969
- [Background] The University of Iowa Otolaryngology Protocols. https://medicine.uiowa.edu/iowaprotocols/maximum-recommended-doses-andduration-local-anesthetics
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343